CLINICAL TRIAL: NCT06404450
Title: Transforming Health and Reducing PerInatal Anxiety Through Virtual Engagement (the HOPE THRIVE STUDY)
Brief Title: Transforming Health and Reducing Perinatal Anxiety Through Virtual Engagement
Acronym: THRIVE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The trial has experienced accrual difficulties and is halted pending additional funding for study recruitment and operations.
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Illinois at Urbana-Champaign (Other); Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other); California State University, Northridge (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A140673 Ref# 22-10528
Record Dates: First submitted 2024-05-03; First posted 2024-05-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital cognitive behavioral therapy (dCBT) (Experimental): The experimental group participants will receive "immediate" access to the Daylight program.
  Interventions: Behavioral: Digital CBT
- Waitlist Control (No Intervention): The waitlist control group participants do not have access to the Daylight program during the study, which lasts from pregnancy to 8-weeks after delivery. However, they will be given access to Daylight after completing the 10-week follow-up survey.

INTERVENTIONS:
Behavioral: Digital CBT — The digital CBT program is called Daylight (Big Health, Ltd). The program employs a virtual therapist to guide individuals through interactive exercises and animations to facilitate the learning and implementation of CBT techniques. The program focuses on four modules (10-20 minutes each) which address specific CBT principles: stimulus control, applied relaxation, cognitive restructuring (decatastrophizing), and imaginal exposure. Daylight is designed to be self-paced, with the app encouraging users to practice techniques both within the app and in real-life situations on a daily basis. Users receive reminders and motivational messages via emails, push notifications, and text messages tailored to participant progress.
  Other Names: Daylight
  Arms: Digital cognitive behavioral therapy (dCBT)

SUMMARY:
The goal of this clinical trial is to evaluate whether digital cognitive behavioral therapy (dCBT) can be used to address clinical anxiety in marginalized and low-income pregnant people in California. The main question it aims to answer is:

What is the efficacy of digital cognitive behavioral therapy (dCBTI) for reducing clinical anxiety among marginalized and low-income pregnant people?

Participants will receive digital cognitive behavioral therapy immediately, or 10 weeks after enrollment (i.e., waitlist control). Participants will complete surveys and interviews until 6-8 weeks postpartum.

DETAILED DESCRIPTION:
Although therapist-delivered cognitive behavioral therapy (CBT) has been shown to be effective for treating clinical anxiety in non-marginalized pregnant populations, barriers to access exist among pregnant people (e.g., long waitlists, childcare issues, limited appointment windows). Recent innovations have focused on addressing barriers to CBT by adapting it for automated, digital delivery. Digital CBT (dCBT) has been shown to be effective for treating clinical anxiety in mostly White, higher socioeconomic status, pregnant, and non-pregnant populations. Person-centered adaptations of dCBT are likely needed to maximize access in marginalized and low-income pregnant people. This study addresses the critical need to evaluate whether dCBT can be used to address clinical anxiety in marginalized and low-income pregnant people in California.

ELIGIBILITY:
Inclusion Criteria:

* California MediCal participant
* Pregnant, 8-27 weeks gestation by ultrasound
* 18-years of age or older
* English speaking
* 9th grade level of education or more
* Daily access to web-enabled computer, smart phone, or tablet
* Current elevated anxiety symptoms (score on the seven item Generalized Anxiety Disorder (GAD-7)questionnaire of 10 or more

Exclusion Criteria:

* Received CBT for anxiety in the last 12-months
* New or changed dose of prescription medication for anxiety, depressive symptoms, or poor sleep in < 4weeks
* Self-reported diagnosis of schizophrenia, psychosis, bipolar disorder, seizure disorder, substance use disorder, severe cognitive impairment (characterized by experiences like forgetting events, having decreased periods of alertness, decreased social awareness)
* Recent trauma to the head or brain damage
* Serious physical health concerns necessitating surgery or hospitalization in the last 6-months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-07-16 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Anxiety Symptoms | Baseline to 3, 6, and 10-weeks after the program start, and Baseline to 6-8 weeks postpartum
  as measured by the Generalized Anxiety Disorder-7 (GAD-7) after 3-weeks, 6-weeks, and 10- weeks after enrollment, and at 6 to 8 weeks postpartum. The GAD-7 utilizes a sum score and the total score can range from 0-21, with higher scores indicating greater anxiety severity.

SECONDARY OUTCOMES:
Pregnancy- Related Anxiety | Baseline to 3, 6, and 10-weeks after the program start, and Baseline to 6-8 weeks postpartum
  as measured by the Pregnancy Related Anxiety Scale (PRAS) after 3-weeks, 6-weeks, and 10-weeks after enrollment, and at 6 to 8 weeks postpartum. The PRAS utilizes a sum score and the total score can range from 4 to 40, with higher scores indicating more pregnancy-specific anxiety.
Stress Symptoms | Baseline to 3, 6, and 10-weeks after the program start, and Baseline to 6-8 weeks postpartum
  as measured by the Perceived Stress Scale (PSS) after 3-weeks, 6-weeks, and 10-weeks after enrollment, and at 6 to 8 weeks postpartum.The PSS utilizes a sum score and total scores can range from 0-40, with higher scores indicating greater perceived stress.
Depressive Symptoms | Baseline to 3, 6, and 10-weeks after the program start, and Baseline to 6-8 weeks postpartum
  as measured by the Patient Health Questionnaire-9 (PHQ-9) after 3-weeks, 6-weeks, and 10-weeks after enrollment, and at 6 to 8 weeks postpartum. The PHQ-9 utilizes a sum score and total scores can range from 0-27, with higher scores indicating greater depression severity.
Insomnia Symptoms | Baseline to 3, 6, and 10-weeks after the program start, and Baseline to 6-8 weeks postpartum
  as measured by the Insomnia Severity Index (ISI) after 3-weeks, 6-weeks, and 10-weeks after enrollment, and at 6 to 8 weeks postpartum. The ISI utilizes a sum score and total scores can range from 0-28, with higher scores indicating greater insomnia severity.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Jelliffe Pawlowski, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ponting C, Baer RJ, Blackman K, Blebu B, Felder JN, Oltman S, Tabb KM, Jelliffe Pawlowski L. Transforming Health and Reducing Perinatal Anxiety Through Virtual Engagement: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 May 30;14:e70627. doi: 10.2196/70627. PMID 40446294